CLINICAL TRIAL: NCT02502136
Title: The Assessment of Differences in Clinical Safety and Efficacy of Carbon Dioxide Insufflation During Sedated and Conventional Endoscopy
Brief Title: Efficacy and Safety of Carbon Dioxide Insufflation During Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 99-4160A3
Record Dates: First submitted 2015-07-01; First posted 2015-07-20 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-04

CONDITIONS: Carbon Dioxide Insufflation During Colonoscopy
Keywords: CO2 insufflation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- CO2 in sedated colonoscopy (Experimental): Carbon dioxide insufflation during colonoscopy with sedation
  Interventions: Procedure: carbon dioxide insufflation during endoscopy
- Air in sedated colonoscopy (Placebo Comparator): Room air insufflation during colonoscopy with sedation
  Interventions: Procedure: Room air insufflation during endoscopy (Placebo)
- CO2 in mild sedated colonoscopy (Experimental): Carbon dioxide insufflation during colonoscopy with mild sedation
  Interventions: Procedure: carbon dioxide insufflation during endoscopy
- Air in deep sedated colonoscopy (Placebo Comparator): Room air insufflation during colonoscopy with deep sedation
  Interventions: Procedure: Room air insufflation during endoscopy (Placebo)
- CO2 in sedated panendoscopy (Experimental): Carbon dioxide insufflation during panendoscopy with sedation
  Interventions: Procedure: carbon dioxide insufflation during endoscopy
- Air in sedated panendoscopy (Placebo Comparator): Room air insufflation during panendoscopy with sedation
  Interventions: Procedure: Room air insufflation during endoscopy (Placebo)
- CO2 in mild sedated panendoscopy (Experimental): Carbon dioxide insufflation during panendoscopy with mild sedation
  Interventions: Procedure: carbon dioxide insufflation during endoscopy
- Air in deep sedated panendoscopy (Placebo Comparator): Room air insufflation during panendoscopy with deep sedation
  Interventions: Procedure: Room air insufflation during endoscopy (Placebo)

INTERVENTIONS:
Procedure: carbon dioxide insufflation during endoscopy — Efficacy and safety study of carbon dioxide insufflation instead of air during sedated endoscopy
  Arms: CO2 in mild sedated colonoscopy; CO2 in mild sedated panendoscopy; CO2 in sedated colonoscopy; CO2 in sedated panendoscopy
Procedure: Room air insufflation during endoscopy (Placebo) — Efficacy and safety study of carbon dioxide insufflation instead of air during sedated endoscopy
  Arms: Air in deep sedated colonoscopy; Air in deep sedated panendoscopy; Air in sedated colonoscopy; Air in sedated panendoscopy

SUMMARY:
The purpose of this study is to assess the differences of safety and efficacy of carbon dioxide insufflation instead of air during sedated or unsedated endoscopy.

DETAILED DESCRIPTION:
Total 640 participants who are indicated to accept endoscopic examinations or procedures will be enrolled in this study. The participants will be divided into 2 groups according to the examination field, esophagogastroduodenoscopy group (320 participants) and colonoscope group (320 participants). The participants in each group will be divided into sedated endoscope subgroup and sedated and unsedated endoscope subgroup (each subgroup is inclusive of 160 participants). Carbon dioxide (CO2) or room air will be used randomly to insufflate the bowel lumen during the procedure in each subgroup.

ELIGIBILITY:
Inclusion Criteria:

* outpatients referred for panendoscopy or colonoscopy examination

Exclusion Criteria:

* pregnancy, breast feeding, severe chronic obstructive lung disease or severe heart failure, renal function impairment, inability to understand participant information, a history of abdominal surgery, or refusal to participate in this study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2011-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
the participants' discomfort scale after endoscopy | within 24hours

CONTACTS AND LOCATIONS:
Overall Officials: Shuo-Wei Chen, MD, Principal Investigator — Chang Gung Memorial Hospital